CLINICAL TRIAL: NCT03284775
Title: Intraoperative Ultrasound in Patients Undergoing Transsphenoidal Surgery for Pituitary Adenoma: a Prospective Devleopment Study
Brief Title: Intraoperative Ultrasound in Patients Undergoing Transsphenoidal Surgery for Pituitary Adenoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17/0310
Record Dates: First submitted 2017-09-12; First posted 2017-09-15 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intraoperative ultrasound — Patients will undergo transsphenoidal surgery in the usual manner except that an intraoperative ultrasound device will be available for use to better visualise the tumour and surrounding neurovascular structures.

SUMMARY:
Pituitary adenoma can be difficult to cure with approximately a third of patients in contemporary series' undergoing incomplete resection. Over the last decade or so a handful of groups have described the use intraoperative ultrasound to improve resection. Although limited, these proof-of-concept studies suggest intraoperative ultrasound is a safe and effective technological adjunct to transsphenoidal surgery for pituitary adenoma.

In this prospective development study 30 adult patients will undergo transsphenoidal surgery for pituitary adenoma with prototype intraoperative ultrasound devices. The primary outcomes will be technical feasibility and device safety. The secondary outcomes will be complete versus incomplete radiological resection, endocrinological remission, the occurrence of postoperative complications, operating time, and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* undergoing transsphenoidal surgery
* diagnosis of pituitary adenoma on pre-operative MRI
* able to provide consent

Exclusion Criteria:

* patients less than 18 years of age
* patients undergoing transcranial surgery
* diagnosis other than that of pituitary adenoma on pre-operative MRI e.g., meningioma
* unable to provide consent e.g., mental illness or later withdrawing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Technical feasibility | Intraoperative
  Technical feasibility will be assessed by the capacity of our system to provide ultrasound images of pituitary and adenoma tissue that correspond to pre- and post-operative MRI.
Device safety | Intraoperative
  Device safety will be assessed by the number, type, and severity of adverse events related to use of the device e.g., device malfunction.

SECONDARY OUTCOMES:
Radiological resection | Early post-operative
  Radiological resection will be determined by a radiologist as gross total resection (GTR), subtotal resection (STR) when more than 80% of the tumour is resected, and partial resection when less than 80% of the tumour is resected.10 Residual tumour will be classified according to its location as intrasellar, suprasellar, intracavernous, or combined.
Endocrinological remission | Early post-operative
  Endocrinological remission will be determined by an endocrinologist. The criteria for acromegaly control will be normalisation of serum insulin-like growth factor and suppression of the nadir serum growth hormone level after oral glucose tolerance test. The criteria for Cushing's disease control will be normalisation of early morning serum cortisol and suppression of serum cortisol after low dose dexamethasone suppression test. The criteria for prolactinoma control will be normalisation of serum prolactin.
Postoperative complications | Early post-operative
  Postoperative complications will include death, cerebrospinal fluid leak, meningitis, vascular complications, visual complications, diabetes insipidus transient and permanent, hypopituitarism, and cranial nerve injury. Vascular complications will include carotid or other vessel injury, or symptomatic haematoma. Venous bleeding from the cavernous sinus will be considered a vascular complication only if it prevents completion of the surgical procedure. Epistaxis will only be considered a vascular complication if it warrants return to the operating room. Cerebrospinal fluid leaks will include all postoperative leaks, and all patients who develop an intraoperative leak requiring lumbar drainage. Patients with Cushing's disease receiving postoperative cortisol, or in whom a hypophysectomy was carried out will also not be included as surgical complications.
Operating time (minutes) | Intra-operative
Length of stay (days) | Early post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital for Neurology and Neurosurgery, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No